CLINICAL TRIAL: NCT02077634
Title: Randomized Phase-II Trial of Abiraterone Acetate Plus LHRH-therapy Versus Abiraterone Acetate Sparing LHRH-therapy in Patients With Progressive Chemotherapy-naïve Castration-resistant Prostate Cancer (SPARE)
Brief Title: Trial of Abiraterone Acetate Plus LHRH-therapy Versus Abiraterone Acetate Sparing LHRH-therapy in Patients With Progressive Chemotherapy-naïve Castration-resistant Prostate Cancer (SPARE)
Acronym: SPARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPARE-001; AUO study number (Other: AP 67/11)
Record Dates: First submitted 2013-12-09; First posted 2014-03-04 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- abiraterone acetate + prednisone + LHRH-therapy (Active Comparator): Patients randomized to this group will continue their LHRH-therapy.
  Interventions: Drug: abiraterone acetate + prednisone + LHRH-therapy
- abiraterone acetate + prednisone (Active Comparator): Patients randomized to this group will stop LHRH-therapy.
  Interventions: Drug: abiraterone acetate + prednisone

INTERVENTIONS:
Drug: abiraterone acetate + prednisone + LHRH-therapy — Hormon therapy will go on
  Arms: abiraterone acetate + prednisone + LHRH-therapy
Drug: abiraterone acetate + prednisone — ormon therapy will be stopped
  Arms: abiraterone acetate + prednisone

SUMMARY:
This is an exploratory Phase 2 multicenter, randomized, open-label study with a randomization allocation ratio of 1:1 [abiraterone acetate + prednisone + LHRH-therapy (Arm A) versus abiraterone acetate + prednisone (Arm B)]. For both groups patients will receive a dose of 1000 mg abiraterone acetate and 10mg prednisone daily (QD). Study drug will be administered as 4 x 250-mg abiraterone acetate tablets and prednisone will be administered as 5 mg orally twice a day (BID). Patients randomized to the LHRH-therapy group will receive the same LHRH-therapy they received prior to entering the trial. 70 medically castrated male patients with metastatic CRPC who have shown tumor progression and are non- or mildly-symptomatic will be enrolled from approximately 12 German study sites.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Written Data Protection Consent has been obtained
3. Male aged 18 years and above
4. Histologically or cytologically confirmed adenocarcinoma of the prostate
5. Metastatic disease documented by positive CT/MRI and/or bone scan (both must be performed). If lymph node metastasis is the only evidence of metastasis, it must be ≥2 cm in diameter
6. Prostate cancer progression documented by PSA according to PCWG2 or radiographic progression according to modified RECIST criteria
7. Asymptomatic or mildly symptomatic from prostate cancer. A score of 0-1 for the question of worst pain within last 24 hours (Appendix 8) will be considered asymptomatic, and a score of 2-3 will be considered mildly symptomatic.
8. Medically castrated, with testosterone levels of <20-50 ng/dl (< 2.0 nM).
9. Combined androgen blockade is permitted, but not required. If patients received combined androgen blockade with an anti-androgen they must have shown PSA progression after discontinuing the anti-androgen prior to enrollment (≥4 weeks since last flutamide, ≥6 weeks since last bicalutamide or nilutamide).
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2 (Appendix 6)
11. Hemoglobin ≥9.0 g/dL independent of transfusion
12. Platelet count ≥100,000 /μl
13. Serum albumin ≥3.0 g/dl
14. Serum creatinine < 1.5 x ULN or a calculated creatinine clearance ≥60 ml/min (Appendix 7)
15. Serum potassium ≥3.5 mmol/l
16. Liver function:

    1. Serum bilirubin <1.5 x ULN (except for patients with documented Gilbert's disease)
    2. AST or ALT <2.5 x ULN
17. Able to swallow the study drug whole as a tablet
18. Life expectancy of at least 6 months
19. Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator and sponsor during the study and for 1 week after last study drug administration.

Exclusion Criteria:

1. Surgical castration (i.e. orchiectomy).
2. Application of any LHRH-therapy (LHRH-analogue or LHRH-antagonist) within 3 months (for patients receiving a 3-months formulation) or 1 months (for patients receiving a 1-month formulation) prior to Cycle 1 day 1.
3. Patients receiving a 6- or 12-months formulation of LHRH-therapy
4. Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
5. Any chronic medical condition requiring a higher dose of corticosteroid than 5mg prednisone/prednisolone bid.
6. Pathological finding consistent with small cell carcinoma of the prostate
7. Liver or visceral organ metastasis
8. Known brain metastasis
9. Use of opiate analgesics for cancer-related pain, including codeine, tramadol, tilidin and others (see Appendix 9), currently or anytime within 4 weeks of Cycle 1 Day 1.
10. Prior cytotoxic chemotherapy or biologic therapy for the treatment of CRPC
11. Radiation therapy for treatment of the primary tumour within 6 weeks of Cycle 1, Day 1
12. Radiation or radionuclide therapy for treatment of metastatic CRPC
13. Prior treatment with Abiraterone acetate or other CYP17 inhibitors (ketoconazole, TAK700, TOK001) ), Enzalutamide (Xtandi) or investigational agents targeting the androgen receptor for prostate cancer for more than 7 days
14. Prior systemic treatment with an azole drug (e.g. fluconazole, itraconazole) within 4 weeks of Cycle 1, Day 1
15. Prior flutamide (Eulexin) treatment within 4 weeks of Cycle 1, Day 1 (patients whose PSA did not decline for three or more months in response to antiandrogen given as a second line or later intervention will require only a two week washout prior to Cycle 1, Day 1)
16. Bicalutamide (Casodex), nilutamide (Nilandron) within 6 weeks of Cycle 1 Day 1 (patients whose PSA did not decline for three or more months in response to antiandrogen given as a second line or later intervention will require only a two week washout prior to Cycle 1, Day1)
17. Uncontrolled hypertension (systolic BP ≥160 mmHg or diastolic BP ≥95 mmHg). Patients with a history of hypertension are allowed provided that blood pressure is controlled by anti- hypertensive treatment
18. Active or symptomatic viral hepatitis or chronic liver disease
19. History of pituitary or adrenal dysfunction
20. Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease or cardiac ejection fraction measurement of <50 % at baseline
21. Any condition that requires treatment with Digoxin, digitoxin, and other digitalis drugs
22. Atrial Fibrillation, or other cardiac arrhythmia requiring therapy
23. Other malignancy with a ≥30 % probability of recurrence within 24 months, except non- melanoma skin cancer.
24. Administration of an investigational therapy within 30 days of Cycle 1, Day 1
25. Any condition, which, in the opinion of the investigator, would preclude participation in this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
radiographic-progression-free survival | 12 month
  The primary objective of the study is to analyze the clinical benefit of abiraterone acetate plus prednisone while sparing LHRH-therapy in chemotherapy-naïve patients with metastatic castration-resistant prostate cancer (CRPC).

SECONDARY OUTCOMES:
Correlation of radiographic-progression-free survival with early PSA-response | 12 month
  To establish additional clinically relevant information regarding early PSA responses to abiraterone and to correlate these with radiographic-progression free survival
Hormonal analyses | 12 month
  To investigate effects of both treatment arms on hormones of the pituitary gonadal axis
Adverse Events | 12 month
  To characterize the safety profile of abiraterone acetate while sparing LHRH-therapy in comparison to continuing LHRH-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Carsten-Henning Ohlmann, PD Dr., Principal Investigator — University Hospital, Saarland
Locations (22):
- Germany (22):
  - Gemeinschaftspraxis für Onkologie, Augsburg
  - Gemeinschaftspraxis für Urologie, Berlin
  - Urologie Bonn-Rhein-Sieg, Praxis Bad Godesberg, Bonn
  - Praxisgemeinschaft für Urologie, Borken
  - Facharztpraxis Dr. Klier, Cologne-Study-Group, Cologne
  - Urologicum Duisburg, Duisburg
  - Urologicum Hamburg, Hamburg
  - Universitätsklinikum Homburg/Saar, Klinik für Urologie und Kinderurologie, Homburg/Saar
  - Urologische Gemeinschaftspraxis, Kempen
  - Klinikum Landshut, Landshut
  - Urologisches Zentrum Lübeck (UZL), Lübeck
  - Gemeinschaftspraxis PUR-R, Mülheim
  - Gemeinschaftspraxis Urologie Pasing, München
  - Privatärztliche urologische Studienpraxis, Nürtingen
  - Pandamed - Übag, Remscheid
  - Zentrum für Onkologie und Urologie Rostock, Wissenschaftskontor Nord GmbH & Co. KG, Rostock
  - Praxisgemeinschaft für Onkologie und Urologie, Wilhelmshaven
  - Praxisgemeinschaft, Wolfsburg
  - DGU, Wuppertal
  - Pandamed - Übag, Wuppertal
  - Praxis für Urologie, Würselen
  - Praxis für Urologie, Zwickau

REFERENCES:
- [Derived] Ohlmann CH, Jaschke M, Jaehnig P, Krege S, Gschwend J, Rexer H, Stockle M. Abiraterone acetate plus LHRH therapy versus abiraterone acetate while sparing LHRH therapy in patients with progressive, metastatic and chemotherapy-naive, castration-resistant prostate cancer (SPARE): study protocol for a randomized controlled trial. Trials. 2017 Oct 4;18(1):457. doi: 10.1186/s13063-017-2195-x. PMID 28978327